CLINICAL TRIAL: NCT06189014
Title: The International PERForator ANeurysm Registry (PERFAN) - Natural History, Treatment, and Outcome of Intracranial Perforator Aneurysms
Brief Title: The International PERForator ANeurysm Registry (PERFAN)
Acronym: PERFAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-01778
Record Dates: First submitted 2023-12-04; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Aneurysm, Brain
Keywords: Perforator Aneurysm; Natural History; Treatment Options; Outcomes
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this international, multicenter, mixed retrospective-prospective, exploratory, observational study is to establish an international registry to fill the knowledge gap created by the rarity of lenticulostriate and basilar perforator aneurysms and the resulting lack of knowledge about their natural history, diagnostic evaluation, management, and clinical outcomes. Specifically, comparative analyses of outcomes in patients with intracranial perforator aneurysms treated conservatively, endovascularly, and surgically will be performed. The study will also evaluate the size and location of lenticulostriate and basilar intracranial perforator aneurysms, collect information on the specific type of endovascular treatment used, compare patients with predominantly perimesencephalic subarachnoid hemorrhage (SAH) who have a perforator aneurysm to those without, and evaluate spontaneous occlusion in conservatively treated aneurysms. Core lab analysis of these aneurysms on various imaging modalities will be performed at the Inselspital and changes in aneurysm characteristics over time will be documented. In addition, the relationship between baseline characteristics and aneurysm characteristics on the incidence of hemorrhage will be examined. The study will involve approximately 20-30 centers worldwide with an estimated total sample size of 200-300 patients by 2025.

DETAILED DESCRIPTION:
1. Background and current state of research

   Lenticulostriate and basilar perforator aneurysms are extremely rare subtypes of intracranial aneurysms. Recent years have seen an increase in their diagnosis due to advancements in imaging technology. However, their low incidence has left a significant gap in the understanding of their natural history, diagnostic evaluation, management, and clinical outcomes. To date, the available literature consists mainly of case reports or small case series, with only a limited number of systematic reviews, such as those on lenticulostriate aneurysms (112 cases) and basilar perforator aneurysms (54 patients).

   The most common presentation of perforator aneurysms is rupture, although unruptured aneurysms may be diagnosed as an incidental finding or as the cause of compressive symptoms. Initial angiography fails to identify approximately 30%-60% of perforator aneurysms. Various treatment approaches have been reported, including surgery and various endovascular techniques such as coiling, embolization with liquid embolic agents, flow-diverters, and even electrothrombosis with a microguidewire. However, all invasive strategies have inherent periprocedural risks that must be carefully weighed against the reported overall high rate of favorable outcomes in conservatively managed patients.

   Despite the growing interest and knowledge in this field, an international multicenter registry that includes baseline patient characteristics, imaging, follow-up protocols, treatment strategies, and outcomes for both ruptured and unruptured intracranial perforator aneurysms is still lacking.
2. Research questions, hypotheses and aims

   The research questions of this exploratory study are:
   * To conduct a comparative analysis of clinical characteristics and outcomes among patients with intracranial lenticulostriate and basilar perforator aneurysms treated conservatively, endovascularly, and surgically.
   * To assess the size and exact location of lenticulostriate and basilar intracranial perforator aneurysms.
   * To gather information regarding the specific type of endovascular treatment employed.
   * To compare patients with predominantly perimesencephalic SAH harboring a perforator aneurysm and those without an aneurysm.
   * To investigate the occurrence of spontaneous occlusion in aneurysms treated conservatively.
   * To perform a core lab analysis of lenticulostriate and basilar intracranial perforator aneurysms using different imaging modalities, including computed tomography (CT), magnetic resonance imaging (MRI), 2D digital subtraction angiography (DSA), and 3D DSA.
   * To review and document observed changes of lenticulostriate and basilar perforator aneurysms (e.g. size) on follow-up imaging.
   * To examine the association between aneurysm size and the incidence of bleeding.
3. Methods

   3.1 Study population

   This is an international, multicenter, mixed-retrospective-prospective exploratory observational study.

   So far, in Switzerland, the Inselspital, the University Hospital Basel, the University Hospital Lausanne, the Regional Hospital of Lugano and the Cantonal Hospital St. Gallen are participating in this study and have received ethical approval. In addition, since the start of the study in early November 2023, already 15 international centers have expressed their interest in participating. More centers worldwide will be contacted via a distribution list [European Society of Minimally Invasive Neurological Therapy (ESMINT); Society of Neurointerventional Surgery (SNIS)] and invited to participate. The investigators estimate that approximately 20-30 centers worldwide will participate with an estimated total sample size of 200-300 patients by 2025. The analysis will be based on a survey (see below for included data) specifically designed for this study and completed by local neuroradiologists, neurologists or neurosurgeons involved in the management of intracranial perforator aneurysms. The primary treating physician will review the clinical records of patients with intracranial perforator aneurysms treated conservatively, endovascularly, or surgically. Study lead and coordination as well as radiological and statistical analysis will be performed by the team at the Inselspital, Bern, Switzerland.

   3.2 Baseline characteristics, imaging variables, treatment variables, and outcome variables

   Data include:
   * Age, sex, relevant comorbidities such as e.g. hypertension, arteriovenous malformation (AVM), Moya-Moya, initial clinical presentation (incidental vs. hemorrhagic). In case of hemorrhagic presentation the type of bleeding [SAH, perimesencephalic subarachnoid hemorrhage (pmSAH), intraventricular hemorrhage (IVH), or intracerebral hemorrhage (ICH)] will be documented.
   * Type of initial diagnostic modality (CT, MRI, DSA).
   * Perforator aneurysm identified on initial diagnostic modality.
   * Type of treatment (surgical vs. endovascular). In case of endovascular treatment specific type [coiling, n-butyl cyanoacrylate (NBCA), ethylene vinyl alcohol (EVOH), flow-diverter, Electro-coagulation, other].
   * Pre- and post-treatment modified Rankin Scale (mRS).

   Clinical endpoints include:
   * mRS at 3 months after initial diagnosis of an intracranial perforator aneurysm
   * mRS at last follow-up (including time-point of last follow-up after diagnosis)
   * Rupture/re-rupture of the index aneurysm as a time-event outcome

   Safety endpoints include:
   * Death during the acute hospital stay
   * Death up to 90 days (related to the index aneurysm)
   * Ischemic stroke (imaging based)
   * Periprocedural and postprocedural complications in patients submitted to endovascular or surgical treatment.

   Efficacy Endpoint

   • For patients receiving treatment, assessment of aneurysm occlusion after treatment and available follow-ups.

   3.3 Data transfer and storage (Medical-Blocks® and REDCap)

   Imaging data from all external participating centers will be securely transferred via and stored on Medical-Blocks® (https://mb-neuro.medical-blocks.ch). This cloud-based platform for storage, anonymization and exchange of medical images in the neuro field (MB-Neuro) is provided by the Inselspital Bern. The platform provides the necessary interfaces to communicate with other secure and advanced IT environments via various Application Programming Interfaces (APIs). Secure Sockets Layers (SSL) with 256-bit encryption is used, which complies with the regulations of KlinV. (Verordnung über klinische Versuche) Art. 18 and HFV (Humanforschungsverordnung) Art. 5 of the Swiss Ordinance on the Storage of Health-Related Personal Data and Biological Materials. The clinical datasets will be provided in an anonymized fashion (matching the anonymized imaging data) by the physician primarily involved in patient management from the participating centers and entered and stored in REDCap.
4. Sample size and statistical analyses

This is an exploratory study. The investigators estimate that approximately 20-30 centers worldwide will participate with an estimated total sample size of 200-300 patients.

Categorical variables will be presented as numbers and percentages, and continuous variables as medians, interquartile range (IQR). Fisher's exact will be used for categorical and Mann-Whitney U test or Kruskal-Wallis test for continuous variables. Logistic regression results will be displayed as odds ratios (OR) for simple regression or adjusted OR (aOR) for multinomial regression analyses, with their corresponding 95% confidence intervals (CIs). As this is an exploratory study, no conclusions about significance can be drawn. Therefore, a p-value < 0.05 will be interpreted as a trend. All analyses will be performed using established statistic software, including R 4.01 or newer, Python 3.83 or newer, Stata 16 and/or Statistical Package for the Social Sciences (SPSS) 27.00 or newer.

ELIGIBILITY:
Inclusion Criteria:

* Patients from the Inselspital and from participating centers worldwide, who have been diagnosed or will be diagnosed with one or more lenticulostriate, basilar and/or other intracranial perforator aneurysms (starting from January 1st, 2013).
* Patients aged ≥18 years
* Written informed consent

Exclusion Criteria:

* Presence of documented written or verbal refusal.
* Aneurysm arising from the middle cerebral artery trunk which does not incorporate a lenticulostriate artery (Vargas Type 1), as they are not perforator aneurysms by strict definition.
* Aneurysm arising from the basilar artery trunk adjacent to a perforating branch but not involving a perforating artery (Satti Type 1), as they are not perforator aneurysms by strict definition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
mRS at 3 months after initial diagnosis of an intracranial perforator aneurysm | 90 days
mRS at last follow-up (including time-point of last follow-up after diagnosis) | Last follow-up, expected to be on average 2 years
Rupture/re-rupture of the index aneurysm as a time-event outcome | Date of rupture/re-rupture
Death during the acute hospital stay | Until patient discharge, up to 4 weeks
Death up to 90 days (related to the index aneurysm) | 90 days
Number of participants with ischemic stroke (imaging based) | Follow-up, expected to be up to 7 days
Periprocedural and postprocedural complications in patients submitted to endovascular or surgical treatment | Peri-/postprocedural, expected to be up to 24 hours
For patients receiving treatment, assessment of aneurysm occlusion after treatment and available follow-ups | First follow-up, expected to be within 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Dobrocky, PD, MD, Principal Investigator — Institute of Diagnostic and Interventional Neuroradiology, Inselspital Bern; Johannes Kaesmacher, Prof, MD, PhD, Principal Investigator — Institute of Diagnostic and Interventional Neuroradiology, Inselspital Bern; Bettina L. Serrallach, MD, Principal Investigator — Institute of Diagnostic and Interventional Neuroradiology, Inselspital Bern
Locations (1):
- Institute of Diagnostic and Interventional Neuroradiology, Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elsheikh S, Mohlenbruch M, Seker F, Berlis A, Maurer C, Kocer N, Jamous A, Behme D, Taschner C, Urbach H, Meckel S. Flow Diverter Treatment of Ruptured Basilar Artery Perforator Aneurysms : A Multicenter Experience. Clin Neuroradiol. 2022 Sep;32(3):783-789. doi: 10.1007/s00062-021-01133-y. Epub 2022 Jan 20. PMID 35059755
- [Background] Gandhi CD, Gilad R, Patel AB, Haridas A, Bederson JB. Treatment of ruptured lenticulostriate artery aneurysms. J Neurosurg. 2008 Jul;109(1):28-37. doi: 10.3171/JNS/2008/109/7/0028. PMID 18590430
- [Background] Granja MF, Monteiro A, Agnoletto GJ, Jamal S, Sauvageau E, Aghaebrahim A, Hanel R. A systematic review of non-trunk basilar perforator aneurysms: is it worth chasing the small fish? J Neurointerv Surg. 2020 Apr;12(4):412-416. doi: 10.1136/neurintsurg-2019-015311. Epub 2019 Oct 9. PMID 31597686
- [Background] Hinojosa-Gonzalez DE, Ferrigno AS, Martinez HR, Farias JS, Caro-Osorio E, Figueroa-Sanchez JA. Aneurysms of the Lenticulostriate Artery: A Systematic Review. World Neurosurg. 2021 Jan;145:471-479.e10. doi: 10.1016/j.wneu.2020.08.160. Epub 2020 Sep 2. PMID 32889194
- [Background] Lu GD, Zhao LB, Jia ZY, Liu S. Micro-guidewire electrocoagulation for the treatment of intracranial aneurysms that are inaccessible by microcatheterization: a case series and review of the literature. J Neurointerv Surg. 2023 Dec;15(12):1229-1233. doi: 10.1136/jnis-2022-019355. Epub 2022 Oct 25. PMID 36283807
- [Background] Ma H, Zhao R, Fang Y, Li Q, Yang P, Huang Q, Xu Y, Hong B, Liu JM. Endovascular electrothrombosis: A promising alternative for basilar artery perforator aneurysm treatment. Interv Neuroradiol. 2021 Aug;27(4):511-515. doi: 10.1177/1591019920987913. Epub 2021 Jan 12. PMID 33435781
- [Background] Mutlu U, Kortman H, Boukrab I. A giant basilar artery perforator aneurysm. Radiol Case Rep. 2022 Jan 14;17(3):911-913. doi: 10.1016/j.radcr.2021.12.034. eCollection 2022 Mar. PMID 35069959
- [Background] Roccatagliata L, Pileggi M, Cianfoni A, Gralla J. Ruptured lenticulostriate artery aneurysm: a report of a case treated with endovascular embolisation. BMJ Case Rep. 2020 Oct 7;13(10):e236649. doi: 10.1136/bcr-2020-236649. PMID 33028571
- [Background] Shlobin NA, Cantrell DR, Ansari SA, Hurley MC, Shaibani A, Jahromi BS, Potts MB. Conservative Management and Natural History of Ruptured Basilar Perforator Artery Aneurysms: Two Cases and Literature Review. World Neurosurg. 2020 Jun;138:218-222. doi: 10.1016/j.wneu.2020.03.042. Epub 2020 Mar 16. PMID 32194275
- [Background] Vargas J, Walsh K, Turner R, Chaudry I, Turk A, Spiotta A. Lenticulostriate aneurysms: a case series and review of the literature. J Neurointerv Surg. 2015 Mar;7(3):194-201. doi: 10.1136/neurintsurg-2013-010969. Epub 2014 Feb 26. PMID 24574545
- [Background] Wu Y, Li Z, Yang D, Wu T, Chen A, Dai C, Zhu Q. Spontaneous subarachnoid hemorrhage caused by ruptured aneurysm of basilar trunk perforator: a case report and literature review. Chin Neurosurg J. 2022 Jun 10;8(1):14. doi: 10.1186/s41016-022-00281-5. PMID 35681227
- [Background] Young M, Schaible P, Asi K, Schaible K. Ruptured Distal Medial Lenticulostriate Artery Aneurysm Treated With Transcortical-Transventricular Approach. Cureus. 2021 Jul 5;13(7):e16186. doi: 10.7759/cureus.16186. eCollection 2021 Jul. PMID 34367793
- [Background] Kumagawa T, Otani N, Kakei Y, Negishi H, Suma T, Yoshino A. Ruptured Basilar Artery Perforator Aneurysm Definitely Diagnosed with Intraoperative Microsurgical Findings: Case Report and Literature Review. NMC Case Rep J. 2023 Jan 16;10:1-7. doi: 10.2176/jns-nmc.2022-0184. eCollection 2023. PMID 36778213
- [Background] van Gijn J, Rinkel GJ. Subarachnoid haemorrhage: diagnosis, causes and management. Brain. 2001 Feb;124(Pt 2):249-78. doi: 10.1093/brain/124.2.249. PMID 11157554